CLINICAL TRIAL: NCT02196233
Title: A Prospective, Randomized Trial Evaluating the Type of Incision on Outcomes and Patient Satisfaction in the Surgical Treatment of Trigger Finger
Brief Title: Surgical Treatment of Adult Trigger Finger
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Douglas Hutchinson, M.D., University of Utah
Other Study IDs: 60239
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Trigger Finger
Keywords: Trigger Finger; Prospective Clinical Research; Randomized; Questionnaires; Transverse; Longitudinal
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Trigger finger is a condition commonly treated with surgical intervention, yet no specific incision type has been associated with improved or worsened scar quality or outcome. Therefore, the investigators objective is to determine if the incision type may affect the results of operative treatment of trigger finger. Therefore, the goals of this study are as follows:

Primary Objective: To directly compare incision type (transverse vs. longitudinal) for trigger finger release with scar quality and patient satisfaction via a validated scar evaluation scale.

Secondary Objective: To directly compare incision type (transverse vs. longitudinal) for trigger finger release to patient outcome via a validated upper extremity outcome score.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 presenting to the four attending surgeons (Don Coleman, Douglas Hutchinson, Andrew Tyser, Angela Wang) through either the University of Utah Orthopaedic Center or the Veteran Affairs Hospital will be evaluated for possible inclusion into the study
* Patients who fail conservative treatment and elect to proceed with open surgical release of the A1 pulley will be offered the option of being included in the study.

Exclusion Criteria:

* Patients aged less than 18, previous failed surgical A1 pulley release, and patients receiving their care outside of the University of Utah Hospital system or the Veteran Affairs Hospital
* In addition, this study will evaluate trigger finger release; patients receiving treatment for trigger thumb will be excluded

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 18 presenting to the four attending surgeons with Trigger Finger
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Trigger Finger Release with Scar Quality and Patient Satisfaction via a Validated Scar Evaluation Scale | 1 Year Follow-up

SECONDARY OUTCOMES:
Trigger Finger Release to Patient Outcome via a Validated Upper Extremity Outcome Score | 1 Year Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hutchinson, Principal Investigator — Orthopedic Surgery
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Saldana MJ. Trigger digits: diagnosis and treatment. J Am Acad Orthop Surg. 2001 Jul-Aug;9(4):246-52. doi: 10.5435/00124635-200107000-00004. PMID 11476534
- [Background] Ryzewicz M, Wolf JM. Trigger digits: principles, management, and complications. J Hand Surg Am. 2006 Jan;31(1):135-46. doi: 10.1016/j.jhsa.2005.10.013. PMID 16443118
- [Background] Sato ES, Gomes Dos Santos JB, Belloti JC, Albertoni WM, Faloppa F. Treatment of trigger finger: randomized clinical trial comparing the methods of corticosteroid injection, percutaneous release and open surgery. Rheumatology (Oxford). 2012 Jan;51(1):93-9. doi: 10.1093/rheumatology/ker315. Epub 2011 Oct 29. PMID 22039269
- [Background] Stefanich RJ, Peimer CA. Longitudinal incision for trigger finger release. J Hand Surg Am. 1989 Mar;14(2 Pt 1):316-7. doi: 10.1016/0363-5023(89)90030-0. No abstract available. PMID 2703681
- [Background] Turowski GA, Zdankiewicz PD, Thomson JG. The results of surgical treatment of trigger finger. J Hand Surg Am. 1997 Jan;22(1):145-9. doi: 10.1016/S0363-5023(05)80195-9. PMID 9018628
- [Background] Froimson, AI. Tenosynovitis and Tennis Elbow; in Green's Operative Hand Surgery, 3rd Edition.
- [Background] Bonnici AV, Spencer JD. A survey of 'trigger finger' in adults. J Hand Surg Br. 1988 May;13(2):202-3. doi: 10.1016/0266-7681_88_90139-8. PMID 3385301
- [Background] Bell MS. Trigger fingers: A checkmark incision. Can J Plast Surg. 2009 Fall;17(3):e18-9. No abstract available. PMID 20808746
- [Background] Brown E, Genoway KA. Impact of diabetes on outcomes in hand surgery. J Hand Surg Am. 2011 Dec;36(12):2067-72. doi: 10.1016/j.jhsa.2011.10.002. PMID 22123050
- [Background] Koh S, Nakamura S, Hattori T, Hirata H. Trigger digits in diabetes: their incidence and characteristics. J Hand Surg Eur Vol. 2010 May;35(4):302-5. doi: 10.1177/1753193409341103. Epub 2009 Aug 17. PMID 19687073
- [Background] Griggs SM, Weiss AP, Lane LB, Schwenker C, Akelman E, Sachar K. Treatment of trigger finger in patients with diabetes mellitus. J Hand Surg Am. 1995 Sep;20(5):787-9. doi: 10.1016/S0363-5023(05)80432-0. PMID 8522745
- [Background] Lim MH, Lim KK, Rasheed MZ, Narayanan S, Beng-Hoi Tan A. Outcome of open trigger digit release. J Hand Surg Eur Vol. 2007 Aug;32(4):457-9. doi: 10.1016/J.JHSB.2007.02.016. Epub 2007 May 4. PMID 17482325
- [Background] Stahl S, Kanter Y, Karnielli E. Outcome of trigger finger treatment in diabetes. J Diabetes Complications. 1997 Sep-Oct;11(5):287-90. doi: 10.1016/s1056-8727(96)00076-1. PMID 9334911
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] van der Wal MB, Verhaegen PD, Middelkoop E, van Zuijlen PP. A clinimetric overview of scar assessment scales. J Burn Care Res. 2012 Mar-Apr;33(2):e79-87. doi: 10.1097/BCR.0b013e318239f5dd. PMID 22249102